CLINICAL TRIAL: NCT05294627
Title: Validation of the Prostate Cancer Biomarker Stockholm3 for Improved Disease Detection and Classification in the Swiss Population
Brief Title: Validation of the Stockholm3 Test for Detection of Prostate Cancer in the Swiss Population
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Department of Urology, University Hospital Freiburg, Freiburg, Germany (Unknown); Department of Urology, Kantonsspital Graubünden, Chur, Switzerland (Unknown)
Responsible Party: Sponsor
Other Study IDs: Stockholm3
Record Dates: First submitted 2022-03-14; First posted 2022-03-24 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Prostate Cancer; Localized Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples (2x10ml)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Stockholm3 — Stockholm3 test prior to prostate biopsy. Prostate biopsy is preformed irrespective of the Stockholm3 score.

SUMMARY:
The purpose of this study is to collect blood samples to investigate the prognostic performance of the STHLM3 test in a population of Swiss and German men suspected of harbouring prostate cancer based on a combination of elevated PSA levels (e.g. >2.5 ng/ml) and/or pathological digital rectal examination and/or MRI-findings.

ELIGIBILITY:
Inclusion Criteria:

* Planned prostate biopsy due to suspicion of prostate cancer (usually due to a combination of elevated PSA levels [e.g. >2.5 ng/ml] and/or pathological digital rectal examination and/or MRI-findings)
* Written informed consent by the participant

Exclusion Criteria:

* Severe anemia (Hb <60g/l)
* Previously already established diagnosis of prostate cancer.

Ages: 18 Years to 99 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Men with suspicion of prostate cancer (usually due to a combination of elevated PSA levels [e.g. >2.5 ng/ml] and/or pathological digital rectal examination and/or MRI-findings)
Sampling Method: Probability Sample
Enrollment: 380 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Cancer detection | 2020-2022
  Correlation between Stockholm3 and histological diagnosis of prostate cancer

SECONDARY OUTCOMES:
Disease state | 2020-2022
  Correlation between Stockholm3 and clinical disease stage

CONTACTS AND LOCATIONS:
Overall Officials: Ashkan Mortezavi, Principal Investigator — Universitätsspital Basel
Locations (1):
- University Hospital Basel, Urology, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No